CLINICAL TRIAL: NCT07159503
Title: Vortex Intelligence Stone Optimized Removal Versus Percutaneous Nephrolithotomy for Treatment of 2-4cm Renal Stones
Brief Title: VISOR Versus PCNL for Treatment of 2-4cm Renal Stones
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-134
Record Dates: First submitted 2025-08-29; First posted 2025-09-08 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-08

CONDITIONS: Kidney Calculi; Kidney Stones
MeSH Terms: conditions — Kidney Calculi | interventions — Nephrolithotomy, Percutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: VISOR (Experimental): Participants will undergo Vortex Intelligence Stone Optimized Removal.
  Interventions: Procedure: Vortex Intelligence Stone Optimized Removal
- PCNL Group (Active Comparator): Participants undergo standard percutaneous nephrolithotomy (PCNL) for renal stone removal.
  Interventions: Procedure: Percutaneous Nephrolithotomy (PCNL)

INTERVENTIONS:
Procedure: Vortex Intelligence Stone Optimized Removal — Vortex Intelligence Stone Optimized Removal integrates irrigation-suction, pressure monitoring-control, and lithotripsy-stone removal functions, aiming to improve stone clearance efficiency, stabilize intrapelvic pressure, and reduce complications.
  Arms: Experimental: VISOR
Procedure: Percutaneous Nephrolithotomy (PCNL) — A standard PCNL technique will be performed according to institutional practice guidelines.
  Arms: PCNL Group

SUMMARY:
The goal of this clinical trial is to learn if the Vortex Intelligence Stone Optimized Removal (VISOR) works safely and effectively to treat kidney stones that are 2 to 4 centimeters in size in kidney. This study will also look at how VISOR compares to the standard surgery, percutaneous nephrolithotomy (PCNL).

The main questions it aims to answer are:

How many participants are stone-free within 24 hours after surgery?

How many participants are stone-free 1 month after surgery?

What side effects or problems, such as pain, fever, or ureter injury, happen with VISOR compared to PCNL?

Does VISOR help keep kidney pressure stable during surgery?

Researchers will compare VISOR to PCNL to see which treatment works better and is safer.

Participants will:

Be randomly assigned to have surgery with either VISOR or PCNL.

Have imaging tests, such as CT scans or ultrasound, after surgery to check if stones were cleared.

Return for follow-up visits about 2 weeks and 1 month after surgery to check recovery and repeat imaging.

About 170 people will take part in this study at cooperative hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Patients with upper urinary tract calculi, where the maximum diameter of a single calculus or the cumulative diameter of multiple calculi is 2-4 cm
* Age between 18 and 80 years, regardless of gender
* Mentally sound and able to comprehend study details and provide informed consent

Exclusion Criteria:

* Presence of ureteral stricture or history thereof
* Previous open or laparoscopic renal and/or ureteral surgery
* Fever (body temperature ≥ 38℃) due to urinary tract infection or other causes within one week prior to surgery
* Pregnancy, lactation, or menstruation at the time of surgery
* ASA classification > Grade 3, indicating severe systemic disease that contraindicates anesthesia or surgery
* Renal anatomical anomalies such as polycystic kidney, horseshoe kidney, or ectopic kidney
* Coagulation dysfunction (e.g., INR > 1.5 or platelet count < 80 × 10⁹/L)
* Intraoperative failure to successfully place the ureteral access sheath

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2025-04-20 (Actual); Primary Completion 2027-02-20 (Estimated); Study Completion 2027-08-20 (Estimated)

PRIMARY OUTCOMES:
Stone-free rate within 24 hours | 24 hours after surgery
  The percentage of participants whose kidney stones are completely cleared within 24 hours after surgery, as confirmed by CT scan.

SECONDARY OUTCOMES:
Stone-free rate at 1 month | 28 ± 7 days after surgery
  The percentage of participants whose stones are completely cleared at 1 month after surgery, evaluated using CT or ultrasound.
Operative Time | During surgery (Day 0)
  Total time from the beginning to the end of the surgery, measured in minutes.
Postoperative fever | 0-30 days after surgery
  Incidence of participants experiencing a body temperature ≥38°C within 30 days after surgery.
Postoperative ureteral stricture | 28 ± 7 days after surgery
  Occurrence of ureteral narrowing detected by imaging within 1 month after surgery.
Pain assessment (VAS score) | Postoperative Day 0-28
  Participants report their pain using the Visual Analog Scale (VAS) at different time points postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Bohan Wang, MD., Ph.D, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China